CLINICAL TRIAL: NCT04115696
Title: Biodegradable Stent Implantation in Biliary Benign Strictures. Spanish Register.
Brief Title: Biodegradable Stent Implantation in Biliary Benign Strictures.
Acronym: BiELLA
Status: Completed | Type: Observational
Sponsor: Group of Research in Minimally Invasive Techniques (Other)
Responsible Party: Sponsor
Other Study IDs: GITMI-03
Record Dates: First submitted 2018-09-12; First posted 2019-10-04 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Biliary Tract; Biliary Tract Diseases; Stenosis; Follow-Up Studies; Stents
MeSH Terms: conditions — Biliary Tract Diseases; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Percutaneous placement of biodegradable biliary stents — The bening biliary strictures stents used in this register are made of polydioxanone (PPDX) (Ella-DV biliary stent, ELLACS, Hradec Králové, Czech Republic). The stents are implanted using a percutaneous transhepatic cholangiography using the standard micropuncture technique. Before stent implantation, balloon bilioplasty may be performed.

SUMMARY:
Spanish registry of resorbable stent implantation in biliary benign strictures.

This registry is sponsored by the Spanish Society of Vascular and Interventional Radiology (SERVEI) and conducted by the Research Group GITMI (Group of Research in Minimally Invasive Techniques) of the University of Zaragoza (Spain).

A software tool hosted on the official website of SERVEI and the journal Intervencionismo will be used for data collection a(https://estudios.watsoncme.com).

DETAILED DESCRIPTION:
This is an prospective observational study of patients that have been implanted a biodegradable stent in the biliary tree.

Patients are recruited when the stent is implanted, and the investigators perfom a patients follow-up during 1, 3, 6, 12, 24, 36, 48 and 52 months.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years-old
* Informed consent
* Non-lithiasic chronic bening single or multiple stenosis
* Possibility of follow-up plus 1 year

Exclusion Criteria:

* Under 18 years old
* Unsigned consent
* Non treatable coagulopathy
* Acute signs of infection
* Diagnosis of neoplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120- 150 patients
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2018-02-03 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Biliary duct patency: bilirubin alterations (> 2.2) | 24 months
  Biliary duct patency after stent implantation evaluating bilirubin alterations
Stent reabsorption: radiographic persistence of stent radiopaque marks | 12 months
  Radiography

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Lozano Blesa Universitary Hospital, Zaragoza, Aragon
  - Hospital Parc Tauli, Sabadell, Barcelona